CLINICAL TRIAL: NCT00363155
Title: Phase I/II Trial of KRN7000 in Patients With Chronic Hepatitis B Infection
Brief Title: KRN7000 in Chronic Hepatitis B
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KRN7000/02-B01
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Hepatitis B, Chronic
Keywords: chronic; hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic; Bronchiolitis Obliterans Syndrome; Hepatitis B | interventions — KRN 7000

INTERVENTIONS:
Drug: KRN7000

SUMMARY:
The purpose of this trial is to determine the safety, tolerability and effectiveness of KRN7000 for chronic hepatitis B infection.

DETAILED DESCRIPTION:
KRN7000 is reported to inhibit HBV replication in HBV transgenic mice. Anti-viral effects of KRN7000 can be expected in HBV, as the compound is able to induce not only IFN-alpha/beta but also IFN-gamma and TNF-alpha. In two clinical trials, KRN7000 was safe in both healthy volunteers and solid cancer patients; particularly, the compound has not been reported to show drug-related serious adverse events. A phase I/II trial is of significance in assessing the safety and efficacy of KRN7000 treatment for CHB patients.

The 300 microgram/m2 dose level, comparable to 10 microgram/kg, can be considered as the highest safe dose level for the phase I/II trial for CHB patients with 3 dose levels. Dose incrementation will be performed in a logarithmic manner: 0.1, 1 and 10 microgram/kg.

In the phase I trial for solid tumor patients, weekly administration of KRN7000 did not allow sufficient time for NKT cell recovery. As KRN7000 is reported to be an activating ligand for NKT cells, it is logical to assume that a dosing interval that provides time for recovery of NKT cells is optimal. In fact, cytokine production after repeating dosing, when NKT cells were hardly detected in the peripheral blood, was not observed. As it took approximately 4 weeks for NKT cells to recover to pre-dose levels after a single administration, monthly administration is now proposed for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (confirmed by a liver biopsy performed within 3 years prior to the screenings visit and HBV DNA in serum >10E5 copies/ml at the screenings visit).
* ALT > 1.2 x ULN on two occasions documented within 8 weeks before initiation of treatment.
* Able and likely to attend regularly for treatment and follow-up.
* Written informed consent.
* Adequate contraception for males and females during treatment and follow-up (written confirmation).

Exclusion Criteria:

* Patients with evidence of cirrhosis.
* Decompensated liver disease, as marked by: bilirubin greater than 20 micromol/L or serum albumin <35 g/L or prothrombin time greater than 3 seconds prolonged or Quick test below 70% or history of bleeding esophageal varices, ascites or hepatic encephalopathy.
* Systemic IFN treatment, systemic antiviral agents, systemic corticosteroids, immune suppressive treatment or any investigational drug within 3 months of entry to this protocol.
* Patients with ALT levels greater than 10 times ULN will not be enrolled but may be followed until three consecutive determinations within 2 months are below this level.
* Pregnancy, or in women of child-bearing potential or in spouses of such women, inability to practice adequate contraception.
* Significant systemic or major illnesses other than liver disease, including congestive heart failure, ischemic heart disease, angina pectoris, cerebrovascular disease, renal failure (creatinine clearance less than 50 ml/min), organ transplantation, serious psychiatric disease or depression, anaphylactic disorder.
* Pre-existing severe cytopenia; Hb<7 mmol/L, WBC <3x10E9/L, Plt <100x10E9/L, Lymphocyte <0.5x10E9/L.
* Any history or presence of autoimmune disease.
* Evidence of hepatocellular carcinoma; alpha-fetoprotein (AFP) levels greater than 50 ng/ml and ultrasound (or other imaging study) within 6 months prior to the entry demonstrating a mass suggestive of liver cancer.
* Human immunodeficiency virus infection, as shown by presence of anti-HIV antibody.
* Patients with cerebroside metabolite abnormalities (e.g. Gaucher's disease).
* Other acquired or inherited causes of liver disease: hepatitis C, hepatitis D, alcoholic liver disease, obesity induced liver disease, drug related liver disease, auto-immune liver disease, Wilson's disease, hemochromatosis, alpha-1-antitrypsin deficiency.
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2003-03; Study Completion 2006-07

PRIMARY OUTCOMES:
To determine safety and tolerability

SECONDARY OUTCOMES:
To evaluate effectiveness in reducing HBV DNA load
To evaluate effectiveness in inducing immunological responses
TO evaluate effectiveness in normalization of ALT

CONTACTS AND LOCATIONS:
Overall Officials: Harry LA Janssen, MD, PhD, Principal Investigator — Dept. of Gastroenterology & Hepatology, Erasmus MC, University Medical Center Rotterdam, Rotterdam, The Netherlands
Locations (1):
- Erasmus MC, University Medical Center Rotterdam, Rotterdam, Netherlands